CLINICAL TRIAL: NCT04124133
Title: Observational Retrospective Study Evaluating Efficacy and Safety of Ialuset Cream or Gauzepad in Second Degree Burns Use for Children
Brief Title: Evaluation of Efficacy and Safety of Ialuset Cream and Gauze in Second-degree Burns on Child
Status: Completed | Type: Observational
Sponsor: Laboratoires Genévrier (Industry)
Responsible Party: Sponsor
Other Study IDs: CHILD study
Record Dates: First submitted 2019-10-10; First posted 2019-10-11 (Actual); Last update posted 2019-10-11 (Actual); Status verified 2019-10

CONDITIONS: Second-degree Burn of Children
MeSH Terms: interventions — Bandages

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: dressing with hyaluronic acid — Application of ialuset cream or gauzepad (hyaluronic acid)

SUMMARY:
Observational retrospective monocentric study occured in the univeristy hospital center of Bensançon the department of pediatric surgery.

Data of patients treated in the hospital between January 2016 and January 2019 have been collected.

DETAILED DESCRIPTION:
Coordinator investigator have put in place a protocol care for children with second degree burns since 2016.

It consists in detersion and cleaning of wound, application of ialuset cream and gauzepad (hyaluronic acid) during 21 days. After 21 days if patients are not healed, physician consider to perform grafting

ELIGIBILITY:
Inclusion Criteria:

* second-degree burns
* less than 20% of the body surface
* less than 15 years old
* treated within 24 hours
* 1st line of treatment with ialuset
* treated at the center between 2016 and 2019

Exclusion Criteria:

* patient who refused data collection

Ages: 1 Month to 15 Years | Sex: All
Age Groups: Child
Study Population: Children from 1month to 15 years with a second degree burn
Sampling Method: Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2018-12-10 (Actual); Primary Completion 2019-04-18 (Actual); Study Completion 2019-04-18 (Actual)

PRIMARY OUTCOMES:
Patient rate with complete healing | 21 days
  pourcentage of patient with 100% of reepithelilisation

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Fotso Kamdem, Principal Investigator — CHU Besançon
Locations (1):
- CHU Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: No